CLINICAL TRIAL: NCT01691924
Title: Randomized, Double Blind, Placebo Controlled "First In-human" Study To Assess the Safety and Tolerability of Single Ascending Oral Doses of PBF-509 in Male Healthy Volunteers
Brief Title: Study To Assess the Safety and Tolerability of PBF-509 in Male Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Palo Biofarma, S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IIBSP-PBF-2012-38
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson Disease
Keywords: Adenosine A2a receptor antagonist; adenosine receptor modulator; Cancer
MeSH Terms: conditions — Parkinson Disease; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules: solid microcrystalline cellulose c.s.p
  Interventions: Drug: Placebo
- PBF-509 (Experimental): The initial dose-escalation scheme includes the following eight doses: 10 mg, 20 mg, 40 mg,80 mg, 160 mg, 320 mg, 480 mg and 620 mg. This dose-escalation scheme has been built with the aim to reach the Minimum Intolerated Dose (MID), i.e. when investigator should stop escalating, and consequently the MTD.
  Interventions: Drug: PBF-509

INTERVENTIONS:
Drug: PBF-509
  Arms: PBF-509
Drug: Placebo
  Arms: Placebo

SUMMARY:
No clinical trials with PBF-509 in humans have been performed to date. Only preclinical studies have been done to assess the pharmacology and pharmacokinetics, the safety and the toxicological profile of the PBF-509.

An initial testing of PBF-509 in humans is planned, starting with the first-into-man clinical trial where a single oral, dose-escalating, and placebo-controlled design will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must meet all of the following inclusion criteria at the pre-study screening visit (within 4 weeks prior to dosing) in order to participate in this study.
* Healthy male subjects, 18-45 years of age.
* Clinically acceptable blood pressure and pulse rate in supine and standing position. Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
* Body weight within normal range (Quetelet's index between 19 and 26) expressed as weight (kg) / height (m2)..
* Non-smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication).
* Able to understand the nature of the study and comply with all their requirements.
* Free acceptance to participate in the study by obtains signed informed consent form approved by the Ethics Committee of the Hospital (CEIC).

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* Background or clinical evidence of chronic diseases.
* Acute illness two weeks before drug administration.
* Having undergone major surgery during the previous 6 months.
* History of alcohol or drug abuse in the last 5 years.
* Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
* Need of any prescription medication within 14 days prior to the administration of the drug and non prescription medication or herbal medicines within 7 days prior to the administration of the drug.
* Participation in other clinical trials during the previous 90 days in which an investigational drug or a commercially available drug was tested.
* Not having donated blood during 3 month period before inclusion in the study.
* Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract.
* 12 lead ECG obtained at screening with PR > 220 msec, QRS>120 msec and QTc >440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG.
* Symptoms of a significant somatic or mental illness in the four week period preceding drug administration.
* History of hepatitis B and / or C and / or positive serology results which indicate the presence of hepatitis B and / or C.
* Positive results from the HIV serology.
* Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation.
* Positive results of the drug screening the day before starting treatment period.
* Known hypersensitivity to the study drug or the composition of the galenical form
* History of psychiatric diseases or epileptic seizures

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 5-7 days post-dose
  Safety and Tolerability evaluation

SECONDARY OUTCOMES:
Pharmacokinetic profile analysis | 0-24 h post dose
  pre-dose; 10; 20; 30; 40; 50; 60; 75 minutes; 1.5h; 2; 2.5; 3; 3.5; 4; 8; 12; 16; 24 hours postdose administration and after recording vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M. Antonijoan, MD, Principal Investigator — Centre de Investigació de Medicaments. Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Palobiofarma S.L. (molecule owner), Mataró, Barcelona
  - Cim- Sant Pau, HSCSP, Barcelona, Catalunya/Barcelona